CLINICAL TRIAL: NCT06137573
Title: A Clinical Study of Absorption, Metabolism and Excretion of [14C]TNP-2198 in Healthy Adult Male Participants- Human Mass Balance and Biotransformation Study of [14C]TNP-2198
Brief Title: Human Mass Balance and Biotransformation Study of [14C]TNP-2198
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TenNor Therapeutics (Suzhou) Limited (Industry)
Responsible Party: Sponsor
Organization: TenNor Therapeutics Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TNP-2198-05
Record Dates: First submitted 2023-11-10; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]TNP-2198 (Experimental): Participants will take a single dose of 600mg 150μCi of [14C]TNP-2198.
  Interventions: Drug: [14C]TNP-2198

INTERVENTIONS:
Drug: [14C]TNP-2198 — 600mg suspension containing 150μCi of [14C] TNP-2198
  Other Names: Rifasutenizol

SUMMARY:
The purpose of the study is to analyze absorption, metabolism, excretion, mass balance and biotransformation after a single oral dose of [14C]TNP-2198 in healthy male participants

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males.
* Age: 18-45 years old (inclusive).
* Body weight: Body mass index (BMI) within 19.0-26.0 kg/m2 (inclusive), and body weight no less than 50 kg.
* Those who have signed the Informed Consent Form voluntarily.
* The participant is able to communicate well with the investigator and to complete the study as specified in the protocol.

Exclusion Criteria:

Those who meet any of the following criteria will not be included:

Auxiliary examinations:

* Those with clinically significant abnormal physical examination, vital signs, clinical laboratory tests (hematology, blood biochemistry, coagulation, urinalysis, and fecal occult blood), thyroid function, 12-lead ECG, chest CT, or abdominal B ultrasonography (liver, gallbladder, pancreas, spleen and kidney).
* Those with positive hepatitis B surface antigen or E antigen, hepatitis C antibody, HIV antibody or syphilis antibody.
* Screening for SARS-CoV-2 infection: clinically significant abnormal C-reactive protein , or positive SARS-CoV-2 nucleic acid.

Medication history:

* Those who have used any drug that inhibits or induces hepatic drug-metabolizing enzymes within 30 days prior to screening.
* Those who have used any prescription drug, over-the-counter drug, Chinese herbal medicine or food supplement, such as vitamins and calcium supplements within 14 days prior to screening.

Medical and surgical history:

* Those with a medical history of any clinically significant disease, or disease or condition that may affect the study results in the opinion of the investigator, including but not limited to the history of cardiovascular system, respiratory system, endocrine system, nervous system, gastrointestinal system, urinary system or hematological, immunological, mental and metabolic diseases.
* Those with a history of organic heart disease, cardiac failure, myocardial infarction, angina pectoris, unexplained arrhythmia, torsade de pointes, ventricular tachycardia, atrioventricular block, prolonged QT syndrome or prolonged QT syndrome symptoms and the family history (confirmed by heredity or sudden death in a close relative at a young age due to cardiac reasons).
* Those who have undergone any major surgery or incompletely healed surgical incision within 6 months prior to screening; major surgery includes, but is not limited to, any surgery with significant risk of haemorrhage, prolonged period of general anesthesia, or incisional biopsy or significant traumatic injury.
* Those with an allergic constitution, such as known history of allergy to two or more substances; or those who may be allergic to the investigational product, or its excipients as judged by the investigator.
* Those with haemorrhoids or perianal disease with regular/ongoing haematochezia, irritable bowel syndrome, or inflammatory bowel disease.

Living habits:

* Those with habitual constipation or diarrhoea.
* Those with alcohol abuse or regular alcohol consumption within 6 months prior to screening, i.e., more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of spirits with 40% alcohol content or 150 mL of wine); or alcohol breath test result ≥ 20 mg/dL at screening.
* Those who smoke more than 5 cigarettes per day or use nicotine-containing products habitually within 3 months prior to screening and are unable to abstain during the study.
* Those who have drug abuse or take soft drugs (such as marijuana) within 3 months prior to screening or take hard drugs (such as cocaine, amphetamines, phencyclidine, etc.) within 1 year prior to screening; or those who have positive urine drug test results at screening.
* Participants who habitually drink grapefruit juice or excessive tea, coffee and/or caffeine-containing beverages, and are unable to abstain during the study.

Others:

* Those who need to work with long-term exposure to radioactive conditions; or those who have significant radiation exposure (≥ 2 chest/abdominal CT scans, or ≥ 3 other X-ray examinations) within 1 year before the study or have participated in radiopharmaceutical labeling trials.
* Those with a history of fear of needles or hemophobia, with difficulty in blood collection or unable to tolerate blood collection by venipuncture.
* Those who have participated in any other clinical trial (including drug and device clinical trials) within 3 months prior to screening.
* Those who have been vaccinated within 1 month prior to screening or plan to be vaccinated during the study.
* Those who plan to have children or donate sperm during the study and within 1 year after the completion of the study, or who do not agree that they and their spouses should take strict contraceptive measures during the study and within 1 year after the completion of the study (see Appendix 3 for details).
* Those who have lost blood or donated 400 mL of blood within 3 months prior to screening or received blood transfusion within 1 month.
* Participants who, in the opinion of the investigator, have any factors unsuitable for participation in this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Cumulative excretion rate of total radioactivity in excreta (urine and feces) | 0 hour(24 hours before administration) to 312 hours after administration. Periodic detection performed, and the collection of biological samples can be judged according to the detection results
  Quantitative analysis of total radioactivity in excreta after oral [14C] TNP-2198 in healthy volunteers
Pharmacokinetics (PK) (AUC0-inf) for TNP-2198 and total radioactivity in plasma and whole blood | 0 hour (60 minutes before administration) to 216 hours after administration. Periodic detection performed, and the collection of biological samples can be judged according to the detection results
  Assessment of pharmacokinetics of TNP-2198 and total radioactivity by measuring the concentration time curve from time zero extrapolated to infinity (AUC0-inf)
PK (AUC0-t) for TNP-2198 and total radioactivity in plasma and whole blood | 0 hour (-60 minutes) before administration to 216 hours after administration. Periodic detection performed, and the collection of biological samples can be judged according to the detection results
  Assessment of pharmacokinetics of TNP-2198 and total radioactivity by measuring the concentration time curve from time zero to the last measureable concentration (AUC0-t)
PK (Cmax ) for TNP-2198 and total radioactivity in plasma and whole blood | 0 hour (60 minutes before administration) to 216 hours after administration. Periodic detection performed, and the collection of biological samples can be judged according to the detection results
  Cmax (maximum observed concentration)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China